CLINICAL TRIAL: NCT00489112
Title: The Use of Medical-Expulsive Therapy With Alfuzocine xl 10mg x1/d for Distal Ureterolithiasis.a Randomized Prospective Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: HaEmek Medical Center, Israel (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 0044-07-EMC
Record Dates: First submitted 2007-06-19; First posted 2007-06-21 (Estimated); Last update posted 2007-06-26 (Estimated); Status verified 2007-06

CONDITIONS: Distal Ureterolithiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Alfuzocine XL 10 mg once a day

SUMMARY:
We will performe a prospective randomized study to evaluate the effects of the addition of alfuzocine xl 10 mg once a day for the conservative treatment of selected ureteral stones. A total of 60 patients with distal ureteral calculi will randomly divide into two treatment groups: group A (n=30) who will receive only analgetic therapy(Dipyrone)and diclofenac i.m. 75mg and group B (n=30) who will receive the same therapy plus alfuzocin xl (10 mg/daily) for a maximum of 2 weeks.No significant differences will be between the groups for age, gender distribution and mean stone size measured in the single largest dimension at presentation.Randomization will be done only with the patients permission after they had read a summary describing the goals of conservative management and a description of the drugs they would be taking. Potential side effects and complications of the drugs were discussed. The expulsion rate will the primary end-point of this study.

ELIGIBILITY:
Inclusion Criteria:

* Stone in the distal ureter until 1 cm of diameter

Exclusion Criteria:

* Evidence of urinary tract infection or sepsis
* Moderate or severe hydronephrosis
* Acute renal failure
* Ureteral stricture
* Stone with >1cm of diameter
* Previuos use of alpha blocker
* Pregnancy
* Previuos ureteral endoscopic or open surgery

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: doron perez, M.D., Principal Investigator — HaEmek MC
Locations (2):
- Israel (2):
  - Haemek medical center,urology department, Afula
  - Haemek Medical Center, Afula